CLINICAL TRIAL: NCT05284370
Title: Modeling of Patient-patient Expert-caregiver Interactions During the Addiction Care Pathway
Brief Title: Interaction Patients Experts During the Addiction Care Pathways
Acronym: IPEXA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200963
Record Dates: First submitted 2022-02-09; First posted 2022-03-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-02

CONDITIONS: Addiction
Keywords: Expert patient; Addictions; Patient engagement; Treatment; Care pathway
MeSH Terms: conditions — Behavior, Addictive; Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"In France and abroad, patient involvement is increasingly encouraged through the development of experiences involving patients in their care or that of their peers.

The Association of PEs in Addictology (APEA) and the Addictology Department of the Bichat Hospital (APHP- Nord, University of Paris) have established a partnership in which PEs volunteer to work with patients throughout the course of their care. To date, no study has evaluated the impact of the PE program in addictology. A preliminary study within the department and the APEA is needed to evaluate the benefits to patients and caregivers, the feasibility and the cost in terms of staff time of implementing the PE program.

The main objective of the project is to describe the care pathways of patients through their interactions with the PEs and the overall addiction care system, over a period of one year, within the Psychiatry-Addictology Department of the Bichat Hospital and then in the outpatient setting.

The secondary objectives are to characterize and describe the patients' profiles according to these pathways; as well as to describe the contribution of EPs in the process of coordinating the care of these patients (interaction between patients - EPs - health professionals).

This is a non-interventional monocentric cohort study in the Psychiatry-Addictology Department of the Bichat Hospital.

In practice, data concerning interactions between patients and EPs and caregivers and EPs will be collected by EPs directly on an eCRF after each contact, for 12 months from inclusion. Patients will be followed during their care pathway for a total of one year, by two telephone assessments at 3 months and 6 months of hospital discharge. A final visit will be made 12 months after hospital discharge by face-to-face interview. Participation will end at the time of the debriefing interview, one year after inclusion.

Modeling the interactions between patients and EPs, and between caregivers and EPs during a course of care in addictology, will lead to a better knowledge of the EP system and the place of EPs in the trajectories of addictology care.

The effectiveness of the PE system can thus be recognized in the management of addictions, in complementarity with the caregivers. The driving factors for implementation will be identified in order to improve the dissemination of the PE system to other centers."

DETAILED DESCRIPTION:
In France and abroad, patient involvement is increasingly encouraged, particularly through the implementation of therapeutic education programs, but also through the promotion of experiences involving patients in their care or that of their peers1 , mainly in the field of chronic diseases and mental health. In this context and for more than 10 years, the Department of Psychiatry - Addictology of the Bichat Hospital has solicited former patients who have developed an expertise, to accompany patients in their addictological care, in addition to the care provided by health professionals.

Over time, their missions have developed considerably and it seemed necessary to integrate them more formally into the care team. It is in this context that the work of formalizing the expert patient system has been carried out, based on existing experiences in France and abroad, particularly in Quebec and Switzerland2,3 . By acting as an intermediary link between patients and caregivers, EPs play a major role in improving the attention paid to patients. They make it possible to put the patient back at the center of care and to give him or her a full place in the care process.

Addictology EPs within the APHP

The APEA and the Addictology Department of the Bichat Hospital (APHP-Nord, University of Paris) have set up a partnership in which expert patients intervene on a voluntary basis with patients throughout the care process, as full partners in care. They are integrated into the care team and, as such, participate in the organization of care and are solicited for service projects.

The clinical missions of the EPs with the patients followed in the service consist, among other things, in co-facilitating the weekly discussion groups with the health professionals, in meeting the hospitalized patients during weekly individual visits and in proposing therapeutic workshops (singing workshop, for example). They are also available before and after hospitalization to maintain the link with the patients they meet, but also to accompany them in the management of their daily life, their emotions and their desire to consume6. Regular exchanges between EPs and caregivers during information meetings allow for better consideration of patients' objectives, desires and plans.

The intervention of expert patients in addictology in the addictology department of the Bichat hospital for the past 10 years has helped fuel the clinical conviction among the care team of the importance of this support in the quality of patient care and in improving their adherence to care. In 2016, the benefits of the EP system, for patients and caregivers alike, were suggested during an evaluation of professional practices (EPP) Finally, as the level of evidence of the PPE was relatively low, it seemed important to think about a larger research project, in order to objectify the nature and impact of EP interventions with patients.

Problem and objectives

The problem is the valorisation of the EP within the care pathway of the addicted patient and the validation of its place as an intermediary link between patients and caregivers in addictology.

Beyond the clinical benefits observed, it is essential that the research results in validated scientific data concerning the fields of action and the place of EPs in the addictology care pathway. This step is essential in order to deploy the EP system in numerous care structures, to allow a larger population to benefit from it, and to enrich the range of therapeutic strategies in addictology.

In the absence of existing data on patient engagement in addictions, a small-scale preliminary study is needed to assess feasibility, time, cost, and risk before conducting a similar project on a larger scale.

In practice, the description of patient-PE and caregiver-PE linkages will constitute a pilot and innovative research project.

The main objective of the project is therefore to describe the care pathways of patients through their interactions with EPs and the overall addiction care system, over a period of one year, within the Psychiatry-Addictology Department of the Bichat Hospital and then in the outpatient setting.

The secondary objectives are to characterize the description of the patients' profiles according to these pathways and to evaluate the coordination of care (interaction between patients - EP - health professionals).

Primary endpoint The main evaluation criterion is the collection and description of the modalities of interaction between EPs and patients.

This description will include the number of contacts, their frequency, duration and modality (group or individual).

These data will be collected by the EPs directly after their interactions with patients and caregivers, on an eCRF.

Secondary endpoint

Patient profile: profile of patients who meet the EPs during their hospitalization in the psychiatry-addictology department of the Bichat hospital to their outpatient care with a one-year follow-up

Data will be collected during their hospitalization and then at 3 months, 6 months and 12 months, by a clinical study technician or the principal investigator, during an individual interview or from the care file:

* The modalities of entry into hospitalization (SAU, hospital consultation, city consultation)
* Post-hospitalization orientation (SSR, psychiatric clinic, addictology outpatient follow-up, psychiatric outpatient follow-up)
* Socio-demographic characteristics
* Addictological history
* Ongoing follow-up / patient-caregiver contact
* Number of re-hospitalizations
* Re-usage/relapse
* Motivation scale
* Professional activity
* Quality of life (scale)
* Compliance with treatment

Care coordination (patient - EP - health professionals interaction):

Care coordination will be assessed via the XXX scale, validated in French, proposed to patients at inclusion and during the end-of-study interview at 12 months.

Exploratory qualitative interviews will be carried out with a representative panel of the different actors of the care pathway (patients, health professionals and EPs) at key moments of the pathway to evaluate the drivers, barriers and evolution of representations (of care, of EPs, of the disease).

Study population Within the Addictology Department of the Bichat site, in 2018, 170 patients with a substance use or addiction disorder were hospitalized without prior exposure to the patient-expert intervention (implemented September 2015). It will be expected that 30% of patients will be lost to follow-up (no care pathway) during the 1-year follow-up. Exploratory analysis using statistical tools such as principal component factor analysis and hierarchical classification will be carried out on 119 care paths.

Patient inclusion criteria

* Adults over 18 years of age, hospitalized during the inclusion period of the study in the addictology department of the Hôpital Bichat-Claude Bernard in Paris
* Substance use disorder, diagnosed according to DSM-5 criteria, i.e. at least 2 diagnostic criteria
* Patients without prior exposure to the PE device
* Patients having received information about the research

Criteria for non-inclusion of patients

* Non comprehension of French
* Patient under guardianship or curatorship
* Patient refusal Criteria for inclusion of health professionals
* Health professionals working in the inpatient unit of the psychiatry-addictology department of the Bichat hospital
* (Or) Health professionals working as outpatients in the psychiatry-addictology department of the Bichat hospital or in outpatient clinics (public, private) and seeing the patients included in the study for follow-up
* Health professionals who received information about the research

Conduct of the research

Patients will be recruited at the time of a full-time hospitalization in the psychiatric addictology unit of the Bichat Hospital.

Data concerning interactions between patients and EPs and caregivers and EPs will be collected by EPs directly on an eCRF after each contact, for 12 months from inclusion.

Patients will be followed during their course of care for a total of one year. Follow-up will be by two telephone assessments at 3 months and 6 months of hospital discharge. Patients will be contacted by phone twice a day, and by SMS, for each visit at D-7, D0 and D+7. If calls are unsuccessful, the patient's referring addictologist (physician or psychologist) and EPs will be contacted for data collection. The patient will be considered lost to follow-up after these three contact methods have failed.

A final visit will be made 12 months after hospital discharge by a face-to-face interview with a clinical study technician or by the principal investigator.

In parallel to the research protocol, the patients will continue their addictological care and their multidisciplinary follow-up, according to the care plan defined during the hospitalization.

Throughout the study, exploratory qualitative interviews will be carried out with a representative panel of the different actors of the care pathway (patients, health professionals and EPs) at key moments of the pathway in order to evaluate the drivers, barriers and evolution of representations (of care, of EPs, of the disease.

Each patient will participate for one year in the study. Participation will end at the time of the review interview with the clinical study technician or principal investigator, one year after inclusion. The inclusion period will be one year. The research may therefore last a total of two years.

This research project will be monocentric, in a single service (recruiting center: Department of Psychiatry and Addictology of the Hôpital Bichat Claude Bernard, hospitalization unit).

ELIGIBILITY:
"Inclusion criteria:

* Adults over 18 years of age, hospitalized during the inclusion period of the study in the addictology department at Hôpital Bichat-Claude Bernard in Paris
* Substance use disorder, diagnosed according to DSM-5 criteria, i.e. at least 2 diagnostic criteria
* Patients without prior exposure to the PE device
* Patients who received information about the research and did not object

Exclusion criteria :

* Non comprehension of French
* Patient under guardianship or curatorship
* Patient under AME
* Patient's refusal".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized full-time for a substance-related disorder or addiction in the Psychiatry-Addictology Department of the Bichat Hospital, exposed for the first time to the patient-expert intervention, followed during one year of addictological care
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Description of patients' care pathways through their interactions with EPs and the overall addiction care system, over a one-year period | Continuously for 1 year
  Description of patients' care pathways through their interactions with EPs and the overall addiction care system, over a one-year period

SECONDARY OUTCOMES:
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  The modalities of entry into hospital (SAU, hospital consultation, city consultation)
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with:
  collaborative practice assessment tool9.
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Post-hospitalization orientation (SSR, psychiatric clinic, addictology outpatient follow-up, psychiatric outpatient follow-up)
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Sociodemographic characteristics - Level of health literacy (Newest Vital SignTM 7 questionnaire)
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Addictological history
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Ongoing follow-up / patient-caregiver contact
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Number of re-hospitalizations
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Re-usage/relapse
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Motivation scale (URICA8)
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Professional activity
Characterize and describe patient profiles according to these pathways | Inclusion, 3 months, 6 months and 12 months
  - Quality of life (EQ-5D-5L scale)
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with: Quality of care delivered,(CACI):
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with: community linkages
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with:empowerment
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with:decision support
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with:care process design
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with: information systems
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with: organization of care.Perceived quality of care(PAT-SAT 3211)
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with: Therapeutic alliance, patient and caregiver (WAI -12 scale)
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with : Continuity of care, as expressed by the patient (Nijmegen Continuity 13)
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with : Patient engagement measured by the Patient Activation Measure.Qualitative evaluation, through sociological, organizational and systemic analysis
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with Stakeholder interviews to identify and describe: The representations of the interviewees on the disease
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with Stakeholder interviews to identify and describe: the care
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with Stakeholder interviews to identify and describe: the PE device
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Evaluation with Stakeholder interviews to identify and describe: the evolution of these representations over time
Describe the contribution of EPs in terms of care coordination (interaction between patients - EPs - health professionals) | During 1 year
  Contextual and organizational elements, drivers or barriers to the implementation and effectiveness of the PE system Potential unexpected effects of EP within the care pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Bichat Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No